CLINICAL TRIAL: NCT02933736
Title: A Phase 0/II Study of Ribociclib (LEE011) in Preoperative Rb-Positive Recurrent High-Grade Glioma and Meningioma Patients Scheduled for Resection to Evaluate Central Nervous System (CNS) Penetration
Brief Title: Ribociclib (LEE011) in Preoperative Glioma and Meningioma Patients
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Nader Sanai (Other)
Collaborators: Novartis (Industry); Ivy Brain Tumor Center (Other); Barrow Neurological Institute (Other)
Responsible Party: Sponsor-Investigator, Nader Sanai, Deputy Director, Ivy Brain Tumor Center, St. Joseph's Hospital and Medical Center, Phoenix
Organization: St. Joseph's Hospital and Medical Center, Phoenix (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PHX-16-0116-80-12
Record Dates: First submitted 2016-10-12; First posted 2016-10-14 (Estimated); Last update posted 2025-03-14 (Actual); Status verified 2025-02

CONDITIONS: Glioblastoma Multiforme; Meningioma
MeSH Terms: conditions — Glioblastoma; Meningioma | interventions — ribociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Administration of ribociclib (Experimental): Subjects will be administered ribociclib prior to surgical resection of their tumor. All patients will be orally-administered 5 doses of LEE011 (900 mg/d) with the final dose occurring at one of 3 following intervals before brain tumor resection:
  Cohort 1: last ribociclib dose 2-4 hours prior to craniotomy for tumor resection
  Cohort 2: last ribociclib dose 6-8 hours prior to craniotomy for tumor resection
  Cohort 3: last ribociclib dose 23-25 hours prior to craniotomy for tumor resection
  Interventions: Drug: Ribociclib

INTERVENTIONS:
Drug: Ribociclib
  Other Names: LEE011

SUMMARY:
In the proposed trial, patients will be administered ribociclib prior to surgical resection of their tumor. Patients will be enrolled in time-intervals sequentially (non-randomized). All patients will be orally-administered 5 doses of LEE011 (900 mg/d) with the final dose occurring at one of 3 intervals before brain tumor resection.

DETAILED DESCRIPTION:
900 mg/d is the maximally tolerated dose (MTD), as determined in a recent Novartis-sponsored Phase I study for advanced solid tumor patients. The recommended dose expansion and Phase 2 is 600mg/d for 3 weeks on and 1 week off. Due to drug pharmacokinetics, the MTD (900mg) dose will be used for pre-surgical dosing in order to maximize the opportunity to identify relevant tumor pharmacokinetic (PK) and pharmacodynamics (PD) endpoints.

To assess the PK, and PD endpoints listed above, cerebrospinal fluid (CSF) and brain tumor tissue will be collected intraoperatively (for gliomas, enhancing and non-enhancing tumor tissue will be collected and analyzed separately). Additionally, blood samples will be obtained at 0.5, 1, 2, 4, 6, 8, and 24 hours after the final ribociclib dose is administered.

Patients with tumors demonstrating positive PK and PD effects will continue treatment with ribociclib (21 days on, 7 days off) after surgery. This will constitute the Phase II component of the study. Patients will be treated until unacceptable toxicity is observed, or until disease progression as assessed by radiographic or clinical metrics. Preliminary rates of progression-free survival in patients with high-grade gliomas and high-grade meningiomas treated with ribociclib will be measured through radiographic and clinical response metrics, specifically Response Assessment in Neuro-Oncology (RANO) criteria and investigator discretion. Overall survival in patients with high-grade gliomas and high-grade meningiomas treated with ribociclib will be assessed by medical record review and survival follow up.

ELIGIBILITY:
Inclusion Criteria

* One prior resection of histologically-diagnosed World Health Organization (WHO) Grade III or IV glioma, or WHO grade II or III meningioma.
* MRI evidence of disease recurrence
* For gliomas, archival tissue must demonstrate: (a) RB positivity on immunohistochemistry OR no RB mutations on next-gen sequencing (NGS), (b) Chromosome 9p21.3 deletion on FISH OR CDKN2A/B/C loss on array CGH OR CDK4/6 or CCND1/2 amplification on array CGH.
* For meningiomas, archival tissue much demonstrate (a) RB positivity on immunohistochemistry OR no RB mutations on next-gen sequencing (NGS).
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2
* Patients ≥ 18 years of age
* Ability to understand and the willingness to sign a written informed consent document (personally or by the legally authorized representative, if applicable).
* Patient has voluntarily agreed to participate by giving written informed consent (personally or via legally-authorized representative(s), and assent if applicable).

(Written informed consent for the protocol must be obtained prior to any screening procedures. If consent cannot be expressed in writing, it must be formally documented and witnessed, ideally via an independent trusted witness.)

* Patients must have recovered from all toxicities related to prior anticancer therapies to ≤ grade 2 (CTCAE v 4.03), provided that concomitant medication is given prior to initiation of treatment with ribociclib. Exception to this criterion: patients with any grade of alopecia are allowed to enter the treatment.
* The following laboratory criteria have been met:

  * Absolute neutrophil count (ANC) ≥1.5 x 109/L
  * Hemoglobin (Hgb) ≥ 9 g/dL
  * Platelets ≥100 x 10^9/L
  * Potassium, total calcium (corrected for serum albumin), magnesium, and sodium within normal limits for the institution or corrected to within normal limits with supplements before first dose of study medication.
  * INR ≤1.5
  * Serum creatinine < 1.5 mg/dL or creatinine clearance ≥ 50 mL/min
  * In the absence of liver metastases, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 2.5 x ULN.
* Serum total bilirubin < ULN, or < 3.0 x ULN in patients with well-documented Gilbert's syndrome.
* Patient with available standard 12-lead ECG with the following parameters at screening (defined as the mean of the ECGs):

  * QTcF interval at screening < 450 msec (using Fridericia's correction)
  * Resting heartrate 50-90 bpm
* Must be able to swallow ribociclib capsules/tablets
* If patient is receiving tamoxifen or toremifene, a washout period of 5 half-lives prior to enrollment is required

Exclusion Criteria:

* Archival tissue not available for research use.
* Archival tumor not Rb-positive status
* No prior radiotherapy
* Co-morbid condition(s) that, at the opinion of the investigator, prevent safe surgical treatment
* Active infection or fever > 38.5°C
* Patients with known hypersensitivity to any of the excipients of ribociclib
* Patients with known hypersensitivity to peanut, soy or lactose
* Prior therapy with ribociclib.
* Patient has a concurrent malignancy or malignancy within 3 years prior to starting study drug, with the exception of adequately treated, basal or squamous cell carcinoma, non-melanomatous skin cancer or curatively resected cervical cancer.
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of the study drugs (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection).
* History of HIV infection (testing not mandatory).
* Other concurrent severe and/or uncontrolled medical condition that would, in the investigator's judgment, cause unacceptable safety risks, contraindicate patient participation in the clinical study or compromise compliance with the protocol.
* Clinically significant, uncontrolled heart disease and/or cardiac repolarization abnormalities.

  * History of acute coronary syndromes (including myocardial infarction, unstable angina, coronary artery bypass grafting, coronary angioplasty, or stenting) or symptomatic pericarditis within 6 months prior to screening
  * History of documented congestive heart failure (New York Heart Association functional classification III-IV)
  * Documented cardiomyopathy
  * Left Ventricular Ejection Fraction (LVEF) <50% as determined by Multiple Gated acquisition (MUGA) scan or echocardiogram (ECHO) at screening
  * Clinically significant cardiac arrhythmias (e.g. ventricular tachycardia), complete left bundle branch block, high-grade AV block (e.g. bifascicular block, Mobitz type II and third-degree AV block)
  * Long QT syndrome or family history of idiopathic sudden death or congenital long QT syndrome, or any of the following:
  * Risk factors for Torsades de Pointe (TdP) including uncorrected hypokalemia or hypomagnesemia, history of cardiac failure, or history of clinically significant/symptomatic bradycardia.
  * Concomitant use of medication(s) with a known risk to prolong the QT interval and/or known to cause Torsades de Pointe that cannot be discontinued (within 5 half-lives or 7 days prior to starting study drug) or replaced by safe alternative medication
  * Inability to determine the QT interval on screening (QTcF, using Fridericia's correction)
  * Systolic blood pressure (SBP) >160 mmHg or <90 mmHg at screening
* Currently receiving any of the following medications and cannot be discontinued 7 days prior to starting study drug:

  * Known strong inducers or inhibitors of CYP3A4/5, including grapefruit, grapefruit hybrids, pomelos/pummelos, star-fruit, pomegranates or pomegranate juice and Seville oranges
  * That have a narrow therapeutic window and are predominantly metabolized through CYP3A4/5
  * Herbal preparations/medications, dietary supplements known as strong inhibitors or inducers of CYP3A4 or those with a known risk of QT prolongation. (Does not include Ca, Mg, Vit D or KCl supplements).
* Currently receiving warfarin or other coumarin-derived anticoagulant for treatment, prophylaxis or otherwise. Therapy with heparin, low molecular weight heparin (LMWH) or fondaparinux is allowed.
* Participation in a prior investigational study within 30 days prior to enrollment or within 5 half-lives of the investigational product, whichever is longer.
* Major surgery within 14 days prior to starting study drug or has not recovered from major side effects (tumor biopsy is not considered as major surgery).
* Has not recovered from all toxicities related to prior anticancer therapies to NCI-CTCAE version 4.03 Grade <1 (Exception to this criterion: patients with grade 1 taxane-induced neuropathy, any grade of alopecia, amenorrhea or other toxicities not considered a safety risk for the patient as per investigator's discretion, are allowed to enter the study.).
* Child-Pugh score B or C.
* History of non-compliance to medical regimen.
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test.]
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing and for 3 months after the last dose of study treatment. Highly effective contraception methods include:

  * Total abstinence (when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
  * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment.
  * Male sterilization (at least 6 months prior to screening) with the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate. For female subjects on the study the vasectomized male partner should be the sole partner for that subject.
  * Use of oral, injected or implanted hormonal methods of contraception or placement of an intrauterine device (IUD) or intrauterine system (IUS), or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception.
  * In case of use of oral contraception, women should have been stable on the same pill for a minimum of 3 months before taking study treatment.
  * Note: Oral contraceptives are allowed but should be used in conjunction with a barrier method of contraception due to unknown effect of drug-drug interaction.
* Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential.
* Sexually active males unless they use a condom during intercourse while taking drug and for 21 days after stopping treatment and should not father a child in this period. A condom is required to be used also by vasectomized men in order to prevent delivery of the drug via seminal fluid.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2016-10-17 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Plasma Exposure | 0.5, 1, 2, 4, 6, 8, and 24 hours post-last 900 mg dosing
CSF Penetration | 2-4, 6-8, and 23-25 hours post-last 900 mg dosing
Brain Accumulation of Ribociclib | Days 1, 22, 43, 64 (add 21 day intervals)...until disease returns or side effect preventing participation in study occurs
  This is the Phase II portion, which assesses trough plasma concentrations of study drug on each clinical visit day, prior to administration of ribociclib on that day.

CONTACTS AND LOCATIONS:
Overall Officials: Nader Sanai, MD, Principal Investigator — Deputy Director of the Ivy Brain Tumor Center
Locations (1):
- Barrow Brain and Spine, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No